CLINICAL TRIAL: NCT07175519
Title: Safety and Efficacy of Aneurysms Treated With Endovascular Devices
Acronym: SEATED
Status: Recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 287395
Record Dates: First submitted 2025-04-15; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-04

CONDITIONS: Brain Aneurysm; Stroke; Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Aneurysm; Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Endovascular treatment of aneurysms — Aneurysm can be treated by endovascular devices using catheters, Treatment modalities can include coils, stents, flow diverters as well as intrasaccular devices

SUMMARY:
In this project the investigators study the safety and efficacy of the recent endovascular devices used in treatment of brain aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing endovascular aneurysm treatment.

Exclusion Criteria:

* All endovascular patients NOT undergoing aneurysm treatment e.g. stents used for stroke treatment; devices and materials used for dAVF, AVM treatments.
* Insufficient background data available e.g., to determine size of aneurysm and device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral aneurysms treated with endovascular devices
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2035-01-15 (Estimated); Study Completion 2035-01-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate predictive factors of aneurysm recurrence after endovascular device embolization (efficacy). | Done at short-term (30 days) post procedural and long term (up to 5 years) post procedural
  Change of aneurysm from Raymond Roy (RR) classification I into RR II or RR III and correlating this with factors such as smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital, London, London, United Kingdom

REFERENCES:
- [Background] Booth TC, Bassiouny A, Lynch J, Sonwalkar H, Bleakley A, Iqbal A, Minett T, Buwanabala J, Narata AP, Patankar T, Islim FI, Kandasamy N, Balasundaram P, Sciacca S, Siddiqui J, Walsh D, Tolias C, Kailaya-Vasan A, Sultan AA, Abd El-Latif M, Mortimer A, Sastry A. Outcome study of the Pipeline Vantage Embolization Device (second version) in unruptured (and ruptured) aneurysms (PEDVU(R) study). J Neurointerv Surg. 2024 Oct 14;16(11):1136-1144. doi: 10.1136/jnis-2023-020754. PMID 38071557